CLINICAL TRIAL: NCT02348840
Title: Mobile Health Intervention to Improve Perinatal Continuum of Care in Guatemala
Brief Title: Perinatal mHealth Intervention in Guatemala
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Gari Clifford, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: IRB00076231; R21HD084114-02 (NIH)
Record Dates: First submitted 2015-01-23; First posted 2015-01-28 (Estimated); Results first posted 2019-08-09 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Pregnancy; Prenatal Care
Keywords: Midwives; Pregnant Women

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- mHealth midwives (Experimental): Midwives will receive access to mHealth technology immediately and use it for 12 months
  Interventions: Device: mHealth
- mHealth midwives - control (Active Comparator): Midwives will not have access to mHealth technology for the first six months, and then will receive the technology for the remaining six months.
  Interventions: Device: mHealth
- Pregnant Women (Active Comparator): Pregnant women may or may not receive mHealth technology, based on the collaborating midwife they are assigned.
  Interventions: Device: mHealth

INTERVENTIONS:
Device: mHealth — A cell phone that can capture data measurements from devices on blood pressure, oxygen level, the heart rate of pregnant women, and the heart rate of the baby.

SUMMARY:
The purpose of the study is to explore ways to improve maternal and child outcomes in the ethnic Maya speaking the Kaqchikel language population, which experiences wide disparities in health care access and outcomes when compared to other inhabitants of Guatemala who are not ethnically Maya and live in other parts of the country.

DETAILED DESCRIPTION:
While advances in medical care have reduced mortality rates across the globe, the same cannot be said for perinatal mortality. This is particularly true of Low and Middle Income Countries (LMICs), which contribute by far the largest proportion of the estimated 5.4 million perinatal deaths annually. Key reasons for this include lack of systematic screening, lack of early health advice-seeking, lack of training for the healthcare workers involved in the healthcare delivery chain and a lack of robust referral. To address these issues, the investigators will introduce and evaluate a scalable mobile health (mHealth) referral system in Guatemala, one of the poorest countries in Latin America with one of the highest perinatal mortality rates. The system combines several key innovations which have been developed over the last 10 years. First, the investigators will introduce a low cost (under $30) ultrasound screening tool, with a blood pressure cuff and pulse oximeter, from which data is fed directly to a smartphone to produce an on-the-spot assessment of the health of the fetus and mother, using a step-by-step pictorial guide (also on the phone). Second, the investigators will implement a mobile phone-mediated medical record and referral system that allows users of both smartphones and basic mobile phones to upload data into a standardized medical record system already in operation in Guatemala. The data will allow healthcare workers to identify or enroll patients, review their histories, and schedule future screenings or follow-up visits, as well as equip the healthcare providers with the necessary information to assess needs, resource allocation and efficacy of treatment or personnel. Thirdly, the investigators will introduce a training protocol for lay midwives to provide routine screening with the system for risk factors such as high blood pressure, fetal growth restriction and fetal distress, and to promote postnatal care coordination. Importantly, this shared system will facilitate communication between the obstetrical care team and the postnatal child care team, which currently represents one of the most pressing care coordination challenges in rural Guatemala. By bringing together engineers, physicians, public health workers, anthropologists, and local nongovernmental organizations to co-design the system around the needs of the existing healthcare infrastructure and the local population, the investigators will create an intuitive system which relieves the burden of data collection, improves diagnostic capabilities, and assists with rapid and accurate referral. The system will also facilitate inter-facility research by introducing a standard medical record protocol.

ELIGIBILITY:
Inclusion Criteria for Midwives:

* Wuqu' Kawoq's catchment area
* Bilingual speakers of Spanish and Kaqchikel Maya
* Willing to give consent and be trained on the mHealth technology
* Must be under the age of 65
* Must be 18 years-old or older

Exclusion Criteria for Midwives:

* Outside Wuqu' Kawoq's catchment area
* Not a bilingual speaker of Spanish and Kaqchikel Maya
* Over the age of 65
* Under the age of 18
* Unable to give consent and be trained on the mHealth technology

Inclusion Criteria for Pregnant Women:

* Must be 18 years-old or older
* Must be pregnant
* Must have a midwife that has been recruited for the study
* Bilingual speakers of Spanish and Kaqchikel Maya
* Willing to give consent

Exclusion criteria for pregnant women

* Under 18 years of age
* Not pregnant
* Does not have a midwife in the study
* Is not bilingual in Spanish and Kaqchikel Maya
* Unable to consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 843 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gari Clifford, PhD, Principal Investigator — Emory University
Locations (1):
- Wuqu' Kawoq, Santiago Sacatepéquez, Guatemala

IPD SHARING:
Plan to Share IPD: Yes
Data will be de-identified and shared through PhysioNet.org. Raw 1-D ultrasound data plus associated demographics will be available.
Supporting Information: Study Protocol, SAP
Time Frame: Data is estimated to become available in 2022 after compilation and analysis is complete.
Access Criteria: Data will be publicly available via PhysioNet.org with no restrictions on analyses.

REFERENCES:
- [Result] Martinez B, Ixen EC, Hall-Clifford R, Juarez M, Miller AC, Francis A, Valderrama CE, Stroux L, Clifford GD, Rohloff P. mHealth intervention to improve the continuum of maternal and perinatal care in rural Guatemala: a pragmatic, randomized controlled feasibility trial. Reprod Health. 2018 Jul 4;15(1):120. doi: 10.1186/s12978-018-0554-z. PMID 29973229
- [Derived] Juarez M, Martinez B, Hall-Clifford R, Clifford G, Rohloff P. Investigating barriers and facilitators to facility-level births in rural Guatemala. Int J Gynaecol Obstet. 2019 Sep;146(3):386-387. doi: 10.1002/ijgo.12865. Epub 2019 Jun 10. No abstract available. PMID 31115904

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Traditional birth attendants (TBAs) were recruited from the municipality of Tecpán Chimaltenango, in rural Guatemala. Enrollment of the TBAs began in January 2015 and eligible pregnant participants were recruited from April 2016 to March 2017. All study follow up ended by February 28, 2018.
Pre-assignment Details: There were 64 TBAs in the study area meeting eligibility criteria who were invited to attend an informational session. Of the eligible TBAs, 49 attended the session and 44 of those individuals agreed to participate in the study.
Groups:
- TBA - Early Access Arm: Traditional birth attendants (TBAs) receiving access to mHealth technology immediately and using it for 12 months
- TBA - Later Access Arm: Traditional birth attendants (TBAs) without access to mHealth technology for the first half of the study who then used mHealth for the remaining time of the 12 month study period
- Pregnant Women - Early Access Arm: Pregnant women under the care of traditional birth attendants in the early access arm
- Pregnant Women - Later Access Arm: Pregnant women under the care of traditional birth attendants in the later access arm
Period: Overall Study
Arm/Group | TBA - Early Access Arm | TBA - Later Access Arm | Pregnant Women - Early Access Arm | Pregnant Women - Later Access Arm
Started | 23 | 21 | 425 | 374
Completed | 21 | 20 | 425 | 374
Not Completed | 2 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes all TBAs and pregnant women for whom demographic data was collected.
Groups:
- Pregnant Women - Early Access Arm: Pregnant women under the care of traditional birth attendants in the early access arm, who completed their pregnancy during the study period
- Pregnant Women - Later Access Arm: Pregnant women under the care of traditional birth attendants in the later access arm, who completed their pregnancy during the study period
- Total: Total of all reporting groups
Arm/Group | TBA - Early Access Arm | TBA - Later Access Arm | Pregnant Women - Early Access Arm | Pregnant Women - Later Access Arm | Total
Number analyzed (Participants) | 23 | 21 | 335 | 327 | 706
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 23 | 21 | 335 | 327 | 706
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 21 | 335 | 327 | 706
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Indigenous Mayan | 23 | 21 | 335 | 327 | 706
Region of Enrollment [Count of Participants; unit: Participants]
  Guatemala | 23 | 21 | 335 | 327 | 706

OUTCOME MEASURES:

1. Primary Outcome: Referral Rates to Local Hospitals
Description: TBAs refer pregnant women to local hospitals for further evaluation or treatment when a pregnancy complications are detected. The median adjusted monthly emergency referral rates (referrals/births) per 100 births for each time period are presented here.
Time Frame: Month 7, Month 12
Population: All TBAs are included in this analysis.
Measure: Median (Inter-Quartile Range); unit: Referrals per 100 births
Groups:
- TBA - Early Access Arm: Traditional birth attendants receiving access to mHealth technology immediately and using it for 12 months
- TBA - Later Access Arm: Traditional birth attendants without access to mHealth technology for the first six months, and then using the technology for the remaining six months
Arm/Group | TBA - Early Access Arm | TBA - Later Access Arm
Number analyzed (Participants) | 23 | 21
Referrals per 100 births
  Month 7 | 33 [22 to 58] | 20 [0 to 30]
  Month 12 | 31 [10 to 42] | 34 [5 to 50]

2. Primary Outcome: Number of Neonatal Deaths
Description: The number of neonatal deaths during the entire study period are presented. Baseline complication rates were unknown for this study population and the study was not powered to detect a difference in the rate of any complication (including neonatal deaths), thus only the total deaths during the entire 12 month period are included.
Time Frame: Month 12
Population: All pregnant participants are included in this analysis.
Measure: Number; unit: deaths
Arm/Group | Pregnant Women - Early Access Arm | Pregnant Women - Later Access Arm
Number analyzed (Participants) | 425 | 374
deaths | 7 | 3

3. Secondary Outcome: Successful Referrals
Description: Referrals to hospitals for further evaluation of possible pregnancy complications were considered to be successful if the pregnant participant went to the hospital after being referred by her TBA. Non-successful referrals were due to the pregnant participant's refusal to go to the hospital (due to lack of permission from a family member, fear, or not recognizing the complication as an emergency) or due to logistical difficulties.
Time Frame: Month 7, Month 12
Population: There were a different number of referrals made during each study period; the overall number analyzed represents the maximum count of referrals in a study period for that study arm.
Measure: Number; unit: Referrals to hospital
Units Other Than Participants: Referrals made during the study period
Arm/Group | TBA - Early Access Arm | TBA - Later Access Arm
Number analyzed (Participants) | 23 | 21
Number analyzed (Referrals made during the study period) | 76 | 51
Referrals to hospital
  First study period: number analyzed (Referrals made during the study period) | 76 | 47
  First study period | 69 | 44
  Second study period: number analyzed (Referrals made during the study period) | 49 | 51
  Second study period | 48 | 47

ADVERSE EVENTS:
Time Frame: Protocol-related adverse events for pregnant participants were collected during the 12 month intervention period.
Description: Only protocol-related serious and non-serious adverse events for pregnant participants were collected. Adverse events were not collected from the traditional birth attendants as adverse events related to the study intervention were not expected to impact these participants.
Arm/Group | TBA - Early Access Arm | TBA - Later Access Arm | Pregnant Women - Early Access Arm | Pregnant Women - Later Access Arm
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 2/425 | 1/374
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/425 | 0/374
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/425 | 0/374

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2014-12-19): https://cdn.clinicaltrials.gov/large-docs/40/NCT02348840/Prot_001.pdf
  • Informed Consent Form (2018-12-05): https://cdn.clinicaltrials.gov/large-docs/40/NCT02348840/ICF_002.pdf